CLINICAL TRIAL: NCT03857256
Title: A Multicenter, Randomized, Double-Blind, Parallel Group, Placebo-Controlled Study To Compare The Efficacy And Safety Of High-Medium Molecular Weight Beta-Glucan As Add-On To Statin Therapy In Subjects With Hyperlipidemia.
Brief Title: Compare the Efficacy and Safety of Beta-Glucan as Add-On to Statin in Subjects With Hyperlipidemia.
Acronym: BetAvena
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Montreal Heart Institute (Other)
Collaborators: Ceapro Inc. (Industry); The Montreal Health Innovations Coordinating Center (MHICC) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PROJ1601
Record Dates: First submitted 2019-02-13; First posted 2019-02-27 (Actual); Results first posted 2024-01-16 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2023-04

CONDITIONS: Hyperlipidemias
MeSH Terms: conditions — Hyperlipidemias | interventions — beta-Glucans

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): matching placebo for 12 weeks.
  Interventions: Drug: Placebo
- Oat beta-glucan 1.5g (Active Comparator): CP105F (Oat beta-glucan) 1.5g (1 tablet of 0.5g TID) for 12 weeks.
  Interventions: Drug: CP105F
- Oat beta-glucan 3g. (Active Comparator): CP105F (Oat beta-glucan) 3g (2 tablets of 0.5g TID) for 12 weeks.
  Interventions: Drug: CP105F
- Oat beta-glucan 6g. (Active Comparator): CP105F (Oat beta-glucan) 6g (4 tablets of 0.5g TID) for 12 weeks.
  Interventions: Drug: CP105F

INTERVENTIONS:
Drug: CP105F — Natural Health Product
  Other Names: beta-glucan
  Arms: Oat beta-glucan 1.5g; Oat beta-glucan 3g.; Oat beta-glucan 6g.
Drug: Placebo — tablet manufactured to mimic the CP105F beta-glucan
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the effects of adding beta-glucan (1.5 g, 3 g or 6 g daily) administered three times a day (TID) in divided doses, to atorvastatin (10 mg - 20 mg) once a day or an equivalent dose of another statin on heart disease lipid risk factors.

DETAILED DESCRIPTION:
Male and female subjects ≥ 18 years of age with an elevated LDL-C > 3.37 mmol/L (130 mg/dL) treated with a stable dose of statin for at least 6 weeks (atorvastatin (10-20mg daily) or equivalent dose of another statin), including subject with previous cardiovascular (CV) events, with partial statin intolerance defined as an inability to tolerate statin therapy in the form and dosages required to achieve treatment goals.

Following signature of informed consent, approximately 264 subjects (66 subjects per beta-glucan treatment group and 22 subjects per matching placebo group) meeting all inclusion criteria and no exclusion criteria will be randomized to receive one of the three doses of beta-glucan (1.5 g, 3 g or 6 g daily) administered TID in divided doses or a matching placebo as an add-on therapy to atorvastatin (10- 20 mg administered once daily) or an equivalent dose of another statin.

The subjects will be assigned to the 3 different doses of beta-glucan or placebo in a tiered fashion as follows:

* The first set of 88 subjects randomized will receive either 1.5 g beta-glucan daily (1 tablet of 500 mg TID) or a matching placebo in a 3:1 ratio,
* The next set of 88 subjects randomized will receive either 3 g of beta-glucan daily (2 tablets of 500 mg TID) or a matching placebo in a 3:1 ratio,
* The last set of 88 subjects randomized will receive either 6 g of beta-glucan daily (4 tablets of 500 mg TID) or a matching placebo in a 3:1 ratio.

During the treatment period, subjects will return to the study site at Visit 3 (Week 6) and at the End of Treatment Visit (Week 12) for laboratory tests and clinical assessments, including Adverse Events (AEs), dietary guidance and study product compliance. At the Safety Follow-up Visit (Week 14), subjects will be contacted via telephone for an assessment of AEs.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet ALL of the following inclusion criteria in order to be eligible for this study:

1. Male or female ≥18 years of age
2. Subjects with hyperlipidemia treated with stable dose of statin for at least 6 weeks; either atorvastatin (10 mg to 20 mg daily) or equivalent dose of another statin at the time of informed consent and with LDL-C level >3.37 mmol/L (130 mg/dL) in fasting conditions at screening
3. Subjects willing to maintain stable standard cholesterol lowering diet (Appendix 2) and physical activity level throughout the study
4. Female of childbearing potential must have a negative urine pregnancy test at screening and randomization baseline Visit 2

   Women are considered not of childbearing potential if they:
   1. Have had a hysterectomy, a bilateral oophorectomy or tubal ligation prior to Combination Therapy Baseline Visit.
   2. Are postmenopausal defined as no menses for at least 1 year and have a serum FSH level of 40 IU/L.

   Women of childbearing potential must agree to use an effective method of birth control throughout the study. Acceptable means of birth control include: implantable contraceptives, injectable contraceptives, oral contraceptives, transdermal contraceptives, intrauterine devices, male or female condoms with spermicide, abstinence, or a sterile sexual partner
5. Ability and willingness to give written informed consent and to comply with the requirements of the study

Exclusion Criteria:

A subject who meets any of the following criteria will NOT be eligible to the study:

1. Use of any other lipid modifying drugs including but not limited to:

   1. Niacin (nicotinic acid) or niacinamide (nicotinamide)
   2. Fibrates or fibric acid derivatives including fenofibrate, gemfibrozil, clofibrate
   3. Bile acid sequestrants including cholestyramine, colesevelam, colestipol
   4. Ezetimibe
   5. PCSK9 inhibitors
   6. Systemic corticosteroids
2. Use of any other lipid modifying supplements within the last 30 days, including but not limited to (a 30-day wash out period is permitted):

   1. Beta-glucan supplements other than the investigational product
   2. Omega-3 fatty acids
   3. Supplements containing flaxseed, fish oil, or algal oil
   4. Sterol/stanol products
   5. Red yeast rice supplements or soy isoflavone supplements
   6. Dietary fiber supplements including > 2 teaspoonful of Metamucil® or psyllium containing supplements per day
   7. Supplements containing oats, oatmeal and oat bran.
3. Use of nonsteroidal anti-inflammatory drugs (NSAIDs) with the exception of acetylsalicylic acid (ASA) at a concentration of up to 325 mg twice a day
4. BMI ≥ 40 kg/m2
5. Female who is pregnant, planning to become pregnant during the study, or breast feeding
6. Subject who is not willing to keep stable the exercise level during the study
7. History of poorly controlled diabetes within the last 3 months (HbA1C >10%)
8. Subjects with poorly controlled blood pressure defined as a sustained mean systolic blood pressure 160 or <100 mmHg and/or diastolic blood pressure 100 or <60 mmHg at screening
9. History of unstable angina, myocardial infarction, coronary artery bypass graft surgery (CABG), percutaneous coronary intervention (PCI), carotid surgery or stenting, cerebrovascular accident, or transient ischemic attack (TIA) within 6 months prior to screening
10. History of heart failure NYHA III-IV within 12 months prior to screening.
11. Subjects with clinically significant electrocardiographic abnormalities
12. Subjects with history of clinically significant endocrine disease known to influence serum lipids
13. Subjects with evidence of hepatic disease (ALT and/or AST greater than 2X ULN, total bilirubin greater than 1.5X ULN, or cirrhosis) at screening
14. Renal dysfunction defined as glomerular filtration rate (GFR) ≤45 mL/min/1.73 m2 at screening
15. Subjects who suffer from inflammatory bowel disease or irritable bowel syndrome
16. Known allergies or intolerance to oats
17. History of malignancy, except subjects who have been disease-free for > 3 yrs or resected basal or squamous cell skin carcinoma or cervical carcinoma in situ
18. Consumption of > 14 alcoholic drinks per week (1 drink = 12 oz beer, 5 oz wine, or 1.5 oz hard liquor at screening). Counseling should be given to encourage the subject to maintain consumption at or below this level throughout the study
19. History of drug abuse
20. Participation in another clinical trial within 30 days of signing the Information and Consent Form (ICF)
21. Any condition or therapy that the investigator believes might pose a risk to the subject or makes participation in the study not in the subject's best interest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2019-05-31 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Claude Tardif, MD, Principal Investigator — Montreal Heart Institute
Locations (1):
- Montreal Heart Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rioux-Labrecque V, Cossette M, Rufiange M, Bilodeau D, Guertin MC, Tardif JC. Supplementation with a beta-glucan tablet has no effect on hyperlipidemia: a randomized, placebo-controlled clinical trial. Am J Clin Nutr. 2023 Jun;117(6):1232-1239. doi: 10.1016/j.ajcnut.2023.04.012. Epub 2023 Apr 11. PMID 37054888

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Oat Beta-glucan 1.5g | Oat Beta-glucan 3g | Oat Beta-glucan 6g
Started | 65 | 66 | 66 | 66
Completed | 64 | 63 | 65 | 63
Not Completed | 1 | 3 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Oat Beta-glucan 1.5g | Oat Beta-glucan 3g | Oat Beta-glucan 6g | Total
Number analyzed (Participants) | 65 | 66 | 66 | 66 | 263
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.7 (9.1) | 59.0 (10.6) | 59.8 (10.7) | 61.7 (9.3) | 59.8 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 39 | 45 | 48 | 169
  Male | 28 | 27 | 21 | 18 | 94
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 2 | 2 | 8
  Not Hispanic or Latino | 63 | 64 | 63 | 64 | 254
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 5 | 3 | 0 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 0 | 2
  White | 62 | 60 | 62 | 66 | 250
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 65 | 66 | 66 | 66 | 263

OUTCOME MEASURES:

1. Primary Outcome: Change in Direct-measured LDL-C
Description: mg/dL
Time Frame: week 0 to week 12
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Placebo | Oat Beta-glucan 1.5g | Oat Beta-glucan 3g. | Oat Beta-glucan 6g.
Number analyzed (Participants) | 65 | 66 | 66 | 66
mg/dL | -3.80 [-13.13 to 5.54] | 2.95 [-2.93 to 8.83] | 4.36 [-3.38 to 12.10] | -1.70 [-8.88 to 5.47]
Statistical Analysis 1: Comparison: Placebo vs Oat Beta-glucan 1.5g vs Oat Beta-glucan 3g. vs Oat Beta-glucan 6g; Tests involving the comparisons of each of the active groups versus placebo for the primary endpoint were conducted at the 0.0167 significance level (to account for three main comparisons); Test type: Superiority — Mean changes from Week 0 in LDL-C were analyzed using a restricted maximum likelihood (REML)-based repeated measures approach including effects of treatment group, time (Week 6 and Week 12) and treatment group x time interaction as well as the covariates of Week 0 value of LDL-C and Week 0 value of LDL-C x time interaction. An unstructured covariance structure were used to model the within-patient errors. Contrasts under this model allowed for the three main comparisons; p = 0.0167, Mixed Models Analysis — Tests involving the comparisons of each of the active groups versus placebo for the primary endpoint were conducted at the 0.0167 significance level (to account for three main comparisons); The Kenward-Roger approximation were used to estimate denominator degrees of freedom

2. Secondary Outcome: Changes in Total Cholesterol,
Description: mmol/L or mg/dL
Time Frame: week 0 to week 12
Reporting Status: Not Posted

3. Secondary Outcome: Changes in Non-High-density Lipoprotein Cholesterol,
Description: mmol/L or mg/dL
Time Frame: week 0 to week 12
Reporting Status: Not Posted

4. Secondary Outcome: Changes in Small Low-density Lipoprotein Subclass Particle Concentration,
Description: nmol/l
Time Frame: week 0 to week 12
Reporting Status: Not Posted

5. Secondary Outcome: Changes in High Sensitivity C-reactive Protein,
Description: mg/L
Time Frame: week 0 to week 12
Reporting Status: Not Posted

6. Secondary Outcome: Changes in Very Low-density Lipoprotein Cholesterol,
Description: mmol/L or mg/dL
Time Frame: week 0 to week 12
Reporting Status: Not Posted

7. Secondary Outcome: Changes in Apo B.
Description: mmol/L
Time Frame: week 0 to week 12
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Changes in HDL-C
Description: mmol/L
Time Frame: week 0 to week 12
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Changes in Triglycerides,
Description: mmol/L
Time Frame: week 0 to week 12
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Changes in Lipoprotein (a) (Lp(a))
Description: mmol/L
Time Frame: week 0 to week 12
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Changes in Glycated Hemoglobin (HbA1c)
Description: percentage
Time Frame: week 0 to week 12
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: The time period covered was from the first dose of IP to safety follow-up visit (week 14).
Arm/Group | Placebo | Oat Beta-glucan 1.5g | Oat Beta-glucan 3g. | Oat Beta-glucan 6g.
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/64 | 0/66 | 0/66
Serious Adverse Events (participants affected / at risk) | 1/65 | 0/64 | 0/66 | 2/66
Other Adverse Events (participants affected / at risk) | 36/65 | 30/64 | 36/66 | 48/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=65) | Oat Beta-glucan 1.5g (N=64) | Oat Beta-glucan 3g. (N=66) | Oat Beta-glucan 6g. (N=66)
Myocardial Infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Transient Ischemic Attack (Nervous system disorders) | 0 | 0 | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=65) | Oat Beta-glucan 1.5g (N=64) | Oat Beta-glucan 3g. (N=66) | Oat Beta-glucan 6g. (N=66)
Flatulence (Gastrointestinal disorders) | 8 | 2 | 6 | 17
Abdominal Distension (Gastrointestinal disorders) | 6 | 2 | 7 | 14
Diarrhoea (Gastrointestinal disorders) | 3 | 2 | 5 | 6
Abdominal Pain (Gastrointestinal disorders) | 3 | 1 | 1 | 1
Abdominal Discomfort (Gastrointestinal disorders) | 1 | 0 | 2 | 7
Constipation (Gastrointestinal disorders) | 2 | 2 | 1 | 1
Faeces soft (Gastrointestinal disorders) | 1 | 0 | 2 | 4
Frequent bowel movements (Gastrointestinal disorders) | 2 | 0 | 0 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3 | 2
Headache (Nervous system disorders) | 3 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 2 | 2 | 0
Herpes Zoster (Infections and infestations) | 0 | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 0 | 2
Abdominal Pain Upper (Gastrointestinal disorders) | 2 | 1 | 0 | 1
Fatigue (General disorders) | 0 | 1 | 2 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Infrequent bowel movements (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Rectal tenesmus (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restriction on the PI is that the sponsor can review material for publication or presentation before public release and can embargo the release for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review. The sponsor can request removal of sponsor's confidential information and the sponsor can request removal of information for which sponsor wishes to obtain intellectual protection.

DOCUMENTS (2):
  • Study Protocol (2020-01-23): https://cdn.clinicaltrials.gov/large-docs/56/NCT03857256/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-14): https://cdn.clinicaltrials.gov/large-docs/56/NCT03857256/SAP_001.pdf